CLINICAL TRIAL: NCT03824990
Title: Multi-center Clinical Study on Early Screening and Treatment of Hyperbilirubinemia of Term and Late-preterm Neonates
Brief Title: Multi-center Clinical Study on Neonatal Hyperbilirubinemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: JiLin Women and Children Health Hospital (Unknown); Shandong Provincial Hospital (Other Government); Shan Dong Qian Fo Shan Hospital (Unknown); Shan Dong Liao Cheng Hospital (Unknown); Guangxi Maternal and Child Health Hospital (Other); Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other); Yin Chuan Maternity and Child Health Hospital (Unknown)
Responsible Party: Principal Investigator, Zhangbin Yu, Nan Jing Maternity and Child Health Care Hospital, Nanjing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NMU-FY2018-72
Record Dates: First submitted 2019-01-30; First posted 2019-01-31 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Quality Improvement; Hyperbilirubinemia, Neonatal
Keywords: Quality improvement; Hyperbilirubinemia; screening; follow-up
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Hyperbilirubinemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Before-intervention phase (No Intervention): All the healthy infants who were admitted from March 2018 to August 2018 to the Well Baby nurse of different hospitals.
- Intervention phase (Experimental): All the healthy infants who were admitted from September 2018 to February 2019 to the Well Baby nurse of different hospitals.During this phase,multiple intervention bundles of quality improvement will be implemented.
  Interventions: Behavioral: Quality improvement of management of neonatal jaundice
- Sustainability intervention phase (Experimental): All the healthy infants who were admitted from March 2019 to August 2019 to the Well Baby nurse of different hospitals.In the Sustainability intervention phase,multiple intervention bundles of quality improvement will be continuous implemented.
  Interventions: Behavioral: Quality improvement of management of neonatal jaundice

INTERVENTIONS:
Behavioral: Quality improvement of management of neonatal jaundice — During the Intervention phase and Sustainability phase ,The hospitals will receive training of multiple evidence based quality improvement methods.
  Arms: Intervention phase; Sustainability intervention phase

SUMMARY:
Eight hospitals in China will participate in the study, which aims to decrease the incidence of severe hyperbilirubinemia.

DETAILED DESCRIPTION:
Through a prospective cohort study of healthy term and near-term infants, the study tries to truly reflect the epidemiology, intervention status, and outcomes of neonatal hyperbilirubinemia and the cost. Hopefully, by improving the quality of management of neonatal jaundice,we can explore and obtain a healthy term and near-term jaundice management model suitable for China's national condition, which can eventually reduce the incidence rate of neonatal severe hyperbilirubinemia and bilirubin encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

term or near-term neonates with gestational age ≥35w and birth weight ≥2000g.

Exclusion Criteria:

Infants admitted to a higher level of intervention before discharge.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20000 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
The incidence of bilirubin encephalopathy | 18 months

SECONDARY OUTCOMES:
The incidence of severe hyperbilirubinemia | 18 months
  Severe hyperbilirubinemia:total serum bilirubin more than 20mg/dL
The rate of lost to follow-up | 18 months
  The rate of lost to follow-up for jaundice after discharge from well-baby nursery
The incidence of adverse neurological outcomes in patients with severe hyperbilirubinemia | 42 months
  Patients with severe hyperbilirubinemia from 11 hospitals will be followed to investigate their neurological outcomes until 24 months after birth
Medical costs in patients with severe hyperbilirubinemia | 18 months
  To compare the medical costs in patients with severe hyperbilirubinemia from 3 phases of quality improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Shuping Han, PHD, Study Director — Nanjing Maternity and Child Health Care Hospital; Zhangbin Yu, PHD, Principal Investigator — Nanjing Maternity and Child Health Care Hospital; Zhiyong Sun, PHD, Principal Investigator — JiLin Women and Children Health Hospital; Haiyan Cai, PHD, Principal Investigator — Qinhuangdao Maternal and Child Health Care Hospital; Yonghui Yu, MD, Principal Investigator — Shandong Provincial Hospital; Xin Yuan, MD, Principal Investigator — Shan Dong Qian Fo Shan Hospital; Jin Qian, MD, Principal Investigator — Shan Dong Liao Cheng Hospital; Jimei Wang, PHD, Principal Investigator — Obstetrics & Gynecology Hospital of Fudan University; Wenyan Tang, PHD, Principal Investigator — Jiangxi Maternal and Child Health Hospital; Qiufen Wei, PHD, Principal Investigator — Guangxi Maternal and Child Health Hospital; Zhankui Li, PHD, Principal Investigator — Northwest Women's and Children's Hospital, Xi'an, Shaanxi; Jie Gu, PHD, Principal Investigator — Yin Chuan Maternity and Child Health Hospital
Locations (1):
- Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu, China